CLINICAL TRIAL: NCT04209764
Title: Prevalenza Del Dolore Nei Dipartimenti di Chirurgia ed Oncoematologia
Brief Title: Prevalence of Pain in the Departments of Surgery and Oncoematology of a Children's Hospital
Status: Completed | Type: Observational
Sponsor: Giuliano Marchetti (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Giuliano Marchetti, Principal Investigator, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Other Study IDs: 1744_OPBG_2019
Record Dates: First submitted 2019-12-16; First posted 2019-12-24 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pain, Postoperative; Chronic Pain Syndrome
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Six years after, the authors will conduct the same analysis to check if there have been any improvements in the management of analgesic therapy after the measures taken according to the results of the previous study conducted in the same departments.

During a single day work three committees, administering a questionnaire to patients or parents, will evaluate the adherence to international recommendations (JCI and WHO) in the management of analgesic therapy.

DETAILED DESCRIPTION:
Thi is a cross sectional study selecting a specific interval (from 8:30 to 17:30) within a single working day of the week, to have a snapshot of the pain experience in a typical working day of the involved departments. The survey will carried out by two pairs of investigators made up of a doctor (possibly Anesthesiologist) and a nurse, not involved in the care of the patient, assigned to hand out a questionnaire-data collection to hospitalized patients or to their parents. Prior informed consent will be obtained by the doctor from parents or from patients more than six years old with the permission of their parents. They will sign a pre-printed paper form specifically formulated for individual ages. For patients and families with inability to understand Italian an interpreter will be used. Only the patients present in the two departments at the time of visit will be included in the study. The two committees will evaluate the adherence to international recommendations (JCI, WHO) in the management of pain treatment, pointing out the prevalence of pain, its intensity and pain therapy prescribed. When necessary, medical records will be consulted in order to verify the "pain history" in the hospital for individual patient and the appropriateness of analgesic administration respecting the intensity of pain experienced. Recorded data will be: 1) patient demographics (age sex, weight, presence of language barriers or cognitive deficits); 2) prevalence and intensity of moderate and/or severe pain during hospitalization, 24 hours before the interview, and at the time of the interview; 3) the type of analgesic administered, the way, the duration and frequency of administration of drugs; 4) the Pain Management Index (PMI) as suggested by Strohbuecker et al and modified for use in children. PMI compares the analgesic drug with the level of pain reported by the patient and is computed by subtracting pain scores from analgesic scores. The analgesics will be scored as follows: no analgesic: 0 points, WHO I: 1 point, WHO II: 2 points, WHO III: 3 points. We defined and scored pain levels of NRS and FLACC 0: no pain (0 points) NRS and FLACC 1-3: mild pain (1 point),.NRS and FLACC 4-6: moderate pain (2 points) and NRS and FLACC 7-10: severe pain (3 points). The PMI ranges from -3 (patients with severe pain receiving no drug at all) to +3 (patients receiving strong opioids and reporting complete pain relief), negative scores indicate undertreatment. For statistical analysis will be used a descriptive analysis using the minimum values, maximum values, averages and standard deviations.

ELIGIBILITY:
Inclusion Criteria:

All the patients in the Ward

Exclusion Criteria:

Patient that are not in the ward at the time of the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Pain in Children: Numbers of patients at the time of interview and twenty four hours before | Forty minutes
  Numbers of patients at the time of interview and twenty four hours before

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano MD Marchetti, Staff, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- BambinoGHRI, Rome, Lazio, Italy

REFERENCES:
- [Derived] Marchetti G, Vittori A, Cascella M, Mascilini I, Piga S, Petrucci E, Castellano A, Caruso R, Francia E, Stocchi F, Marinangeli F, Inserra A, Picardo SG. Pain prevalence and pain management in children and adolescents in an italian third level pediatric hospital: a cross-sectional study. Ital J Pediatr. 2023 Mar 29;49(1):41. doi: 10.1186/s13052-023-01439-2. PMID 36978099